CLINICAL TRIAL: NCT03754972
Title: The Sagittal Plane Shear Index (SPSI) for Planning Whether to Fuse After Decompressing a Stenotic Lumbar Level
Brief Title: Sagittal Plane Shear Index for Planning Lumbar Stenosis Surgery
Acronym: SPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Metrics Diagnostics, Inc (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPSI-01
Record Dates: First submitted 2018-11-14; First posted 2018-11-27 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis; Spondylolisthesis
Keywords: lumbar; spondylolisthesis; instability; diagnosis; treatment planning; fusion; decompression
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Disease

STUDY DESIGN:
Intervention Model Description: Determine whether an objective metric for spinal stability will change the surgical treatment plan in a significant proportion of patients with lumbar spinal stenosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar spinal stenosis surgery candidate (Experimental): Patients with lumbar spinal stenosis and spondylolisthesis that have previously consented to surgical treatment. After recording the initial surgical plan, the Sagittal plane shear index (SPSI) will be provided to the surgeon. The surgeon may change the initial surgical plan based on the stability metric.
  Interventions: Diagnostic Test: Sagittal plane shear index (SPSI)

INTERVENTIONS:
Diagnostic Test: Sagittal plane shear index (SPSI) — Report SPSI to surgeon after surgeon records an initial surgical plan, and determine whether the objective spinal stability metric influences a change in the surgical plan.

SUMMARY:
The objective of the clinical investigation is to assess the proportion of lumbar spinal stenosis surgical treatment plans that change when an objective measurement of spinal stability is included and applied following a simple treatment algorithm. The objective spinal stability metric is calculated from flexion-extension radiographs using previously validated methods.

DETAILED DESCRIPTION:
Patients with previously diagnosed lumbar spinal stenosis and spondylolisthesis, who have consented to surgical treatment consisting of either decompression alone or decompression plus fusion will be invited to participate in the study. The initial surgical plan will be recorded prior to reviewing the sagittal plane shear index (SPSI). The sagittal plane shear index will be calculated flexion-extension radiographs. The measurements required to calculate SPSI will be obtained using previously validated methods. SPSI greater than 2 indicates that the translation-per-degree of rotation (TPDR) is above the upper limit of the 95% confidence interval observed in several hundred asymptomatic and radiographically normal individuals. SPSI will be reported to the surgeon after recording the pre-SPSI surgical plan. The surgeon will then decide whether to change the surgical plan. For example, if the initial surgical plan was to only decompress a level, and SPSI is greater than 2, the surgeon may plan to add fusion to the decompression. Conversely, if the initial plan was decompression plus fusion, and the SPSI indicates that the level is objectively stable, the post-SPSI plan may be to only decompress the level. The proportion of surgical plans that change after reviewing the SPSI report will be determined. If the proportion of surgical plans that change is greater than 15%, further research will be undertaken to explore whether deciding, based on objective measurement of spinal stability, whether to add fusion to decompression of a stenotic lumbar level will have a significant effect on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms consistent with single level lumbar spinal stenosis based on judgment and experience of the investigator
2. Central and or foraminal stenosis confirmed by MRI as per the investigators clinical standards
3. Grades 1 (10 to 25%) or 2 (26 to 50%) anterior or retro-spondylolisthesis using the Meyerding scale [43]
4. Absence of lateral spondylolisthesis
5. No prior lumbar spinal surgery
6. Absence of American Society of Anesthesiologists (ASA) class IV or higher disease
7. The single level surgical technique planned (prior to viewing the spinal motion report) to decompress the level is not expected to destabilize the spine (fusion is not deemed necessary due to probable iatrogenic instability)
8. Prior to viewing the spinal motion report, the surgical plan includes decompression or decompression and fusion of only one level
9. Based on the investigators subjective assessment, the patient is able to flex and extend sufficiently to facilitate acceptable flexion and extension radiographs
10. The fusion technique planned prior to viewing the spinal motion report is the following: Instrumented posterior (pedicle screws and rods) with / without postero-lateral interbody fusion cage
11. Subject is able to understand and sign the study Informed Consent Form
12. Subjects is at least 18 years of age.
13. Subject has willingness and ability to comply with study procedures and visit schedules and able to follow oral and written instructions

Exclusion Criteria:

1. Lumbar stenosis without spondylolisthesis
2. Severe lumbar stenosis that requires a wide decompression where the investigator believes (based on experience and available research studies) that the decompression will destabilize the spine and fusion surgery is required regardless of preoperative SPSI
3. Pregnant women
4. Scoliosis involving a lumbar curve greater than 10 degrees
5. Stenosis at the level of a transitional vertebra
6. Lateral spondylolisthesis (Coronal plane translational misalignment between vertebrae)
7. Prior lumbar spinal surgery
8. American Society of Anesthesiologists (ASA) class IV or higher disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hipp, PhD, Principal Investigator — Medical Metrics Diagnostics, Inc
Locations (3):
- Netherlands (3):
  - OLVG Oost, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided
No current plan to share data from this pilot study

REFERENCES:
- [Background] Staub BN, Holman PJ, Reitman CA, Hipp J. Sagittal plane lumbar intervertebral motion during seated flexion-extension radiographs of 658 asymptomatic nondegenerated levels. J Neurosurg Spine. 2015 Dec;23(6):731-8. doi: 10.3171/2015.3.SPINE14898. Epub 2015 Aug 21. PMID 26296193
- [Background] Rihn JA, Lee JY, Khan M, Ulibarri JA, Tannoury C, Donaldson WF 3rd, Kang JD. Does lumbar facet fluid detected on magnetic resonance imaging correlate with radiographic instability in patients with degenerative lumbar disease? Spine (Phila Pa 1976). 2007 Jun 15;32(14):1555-60. doi: 10.1097/BRS.0b013e318067dc55. PMID 17572627
- [Background] Hipp JA, Guyer RD, Zigler JE, Ohnmeiss DD, Wharton ND. Development of a novel radiographic measure of lumbar instability and validation using the facet fluid sign. Int J Spine Surg. 2015 Jul 17;9:37. doi: 10.14444/2037. eCollection 2015. PMID 26273555
- [Background] Leone A, Guglielmi G, Cassar-Pullicino VN, Bonomo L. Lumbar intervertebral instability: a review. Radiology. 2007 Oct;245(1):62-77. doi: 10.1148/radiol.2451051359. PMID 17885181
- [Background] Zhao K, Yang C, Zhao C, An KN. Assessment of non-invasive intervertebral motion measurements in the lumbar spine. J Biomech. 2005 Sep;38(9):1943-6. doi: 10.1016/j.jbiomech.2004.07.029. PMID 16023484
- [Background] Pearson AM, Spratt KF, Genuario J, McGough W, Kosman K, Lurie J, Sengupta DK. Precision of lumbar intervertebral measurements: does a computer-assisted technique improve reliability? Spine (Phila Pa 1976). 2011 Apr 1;36(7):572-80. doi: 10.1097/BRS.0b013e3181e11c13. PMID 21217439
- [Background] Forsth P, Olafsson G, Carlsson T, Frost A, Borgstrom F, Fritzell P, Ohagen P, Michaelsson K, Sanden B. A Randomized, Controlled Trial of Fusion Surgery for Lumbar Spinal Stenosis. N Engl J Med. 2016 Apr 14;374(15):1413-23. doi: 10.1056/NEJMoa1513721. PMID 27074066
- [Background] Ghogawala Z, Dziura J, Butler WE, Dai F, Terrin N, Magge SN, Coumans JV, Harrington JF, Amin-Hanjani S, Schwartz JS, Sonntag VK, Barker FG 2nd, Benzel EC. Laminectomy plus Fusion versus Laminectomy Alone for Lumbar Spondylolisthesis. N Engl J Med. 2016 Apr 14;374(15):1424-34. doi: 10.1056/NEJMoa1508788. PMID 27074067
- [Background] Machado GC, Ferreira PH, Yoo RI, Harris IA, Pinheiro MB, Koes BW, van Tulder MW, Rzewuska M, Maher CG, Ferreira ML. Surgical options for lumbar spinal stenosis. Cochrane Database Syst Rev. 2016 Nov 1;11(11):CD012421. doi: 10.1002/14651858.CD012421. PMID 27801521
- [Background] Jansson KA, Nemeth G, Granath F, Blomqvist P. Spinal stenosis re-operation rate in Sweden is 11% at 10 years--a national analysis of 9,664 operations. Eur Spine J. 2005 Sep;14(7):659-63. doi: 10.1007/s00586-004-0851-9. Epub 2005 Mar 8. PMID 15754213
- [Background] Tsutsumimoto T, Shimogata M, Yoshimura Y, Misawa H. Union versus nonunion after posterolateral lumbar fusion: a comparison of long-term surgical outcomes in patients with degenerative lumbar spondylolisthesis. Eur Spine J. 2008 Aug;17(8):1107-12. doi: 10.1007/s00586-008-0695-9. Epub 2008 Jun 7. PMID 18536941
- [Background] Eliasberg CD, Kelly MP, Ajiboye RM, SooHoo NF. Complications and Rates of Subsequent Lumbar Surgery Following Lumbar Total Disc Arthroplasty and Lumbar Fusion. Spine (Phila Pa 1976). 2016 Jan;41(2):173-81. doi: 10.1097/BRS.0000000000001180. PMID 26751061
- [Background] Makino T, Kaito T, Fujiwara H, Ishii T, Iwasaki M, Yoshikawa H, Yonenobu K. Does fusion status after posterior lumbar interbody fusion affect patient-based QOL outcomes? An evaluation performed using a patient-based outcome measure. J Orthop Sci. 2014 Sep;19(5):707-12. doi: 10.1007/s00776-014-0591-6. Epub 2014 Jun 12. PMID 24916199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from four tertiary non-academic hospitals in The Netherlands were recruited by employing a non-probability purposive sampling method.
Period: Overall Study
Arm/Group | Lumbar Spinal Stenosis Surgery Candidate
Started | 100
Completed | 75
Not Completed | 25
Not completed — Protocol Violation | 25

BASELINE CHARACTERISTICS:
Groups:
- Lumbar Spinal Stenosis Surgery Candidate: Patients were eligible for participation if they had i) symptoms consistent with single-level LSS, ii) central and/or foraminal stenosis between two adjacent vertebrae confirmed by MRI, iii) grades 1 (10 to 25%) or 2 (26 to 50%) anterior or retro-spondylolisthesis according to the Meyerding classification,28 iv) no history of prior lumbar spinal surgery and v) were suitable for Posterior Lumbar Interbody Fusion (PLIF) surgery using posterior pedicle screws, rods and/or a spinal cage in case instrumented fusion was considered. Patients were excluded if they had i) stenosis at the level of a transitional vertebra or severe stenosis that required a wide decompression that was judged to destabilize the spine, ii) lateral spondylolisthesis, iii) scoliosis involving a lumbar curve > 10 degrees, iv) an American Society of Anesthesiologists (ASA) class IV or higher disease or v) were pregnant.
Arm/Group | Lumbar Spinal Stenosis Surgery Candidate
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.05 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 91
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 100
ODI [Mean (Standard Deviation); unit: units on a scale] | 39.6 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Surgical Plans Recorded Prior to the SPSI Report That Are Altered After Integration of SPSI Into the Surgical Planning
Description: The surgeons will record their surgical plan (decompression alone or decompression plus fusion) prior to receiving the SPSI report. The surgeon will then integrate the data in the SPSI report into their surgical planning and record a post-SPSI report surgical plan. The proportion of lumbar spinal stenosis surgery plans that change after an objective metric for spinal stability is included in the surgical planning will be determined. If the proportion of plans that change after integration of the SPSI report is greater than expected due to subjectivity in surgical planning, then the SPSI report will be considered clinically effective and further research will be pursued.
Time Frame: Pre-surgery
Population: Patients meeting all inclusion criteria, not meeting any exclusion criteria, and where intervertebral rotation at the treatment level was >= 5 degrees between flexion and extension
Measure: Number; unit: Surgical plans
Arm/Group | Lumbar Spinal Stenosis Surgery Candidate
Number analyzed (Participants) | 75
Surgical plans
  SPSI supported surgeons initial surgical plan | 47
  Surgical plan changed after using SPSI in planning | 22
  Surgeons chose not to implament a change in surgical plan supported by the SPSI metric | 6

2. Secondary Outcome: Association Between the Preoperative SPSI and the Facet Fluid Sign Observed in a Preoperative MRI
Description: Prior research has reported that SPSI is significantly higher at lumbar levels where a facet fluid sign is observed in a MRI exam. Outcome 2 is intended to test the hypothesis that this prior finding can be repeated. SPSI will be calculated for all levels in the lumbar spine from preoperative lumbar flexion-extension radiographs. The surgeons will record whether they observe the fluid sign in the facet joints based on review of a preoperative MRI exam. Statistical tests will be performed for an association between preoperative SPSI and the presence or absence of a facet fluid sign observed by the treating surgeon in a preoperative MRI exam of the lumbar spine.
Time Frame: Pre-surgery
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: The Proportion of Surgically Decompressed Levels Where SPSI Was at Least One Standard Deviation Higher at 12 Months Compared to Preoperatively.
Description: Prior research has documented that decompression surgery may compromise the stability of the treated level. To test whether this phenomena can be documented using the SPSI metric, SPSI measured at 12 months will be compared to SPSI measured preoperatively. This will be assessed only in patients treated with decompression alone (patients treated with fusion in addition to decompression will not be included). Statistical tests will be used to determine the proportion of levels treated using decompression only where the SPSI at 12 months was at least 1 standard deviation greater than preoperatively.
Time Frame: One year after surgery
Reporting Status: Not Posted, anticipated posting 2025-09

4. Secondary Outcome: Reoperation Rate at 1 and 2 Years Following Surgery
Description: Multiple prior studies have documented reoperation rates following surgery for lumbar spinal stenosis. To test whether the reoperation rate in the current study is comparable to prior studies, clinical records will be reviewed to determine whether additional surgery was performed at the treated and/or adjacent levels. Statistical tests will be used to compare the reoperation rates at 12 and 24 months after the index surgery to reoperation rates previously reported in the peer-reviewed literature.
Time Frame: 12 and 24 months
Reporting Status: Not Posted, anticipated posting 2025-04

5. Secondary Outcome: Are the ODI Scores at 12 Months Following Lumbar Fusion Surgery Dependent on Whether the Treated Level is Fused, With Fusion Defined as Intervertebral Rotation < 2 Degrees and an Absence of Radiographic Signs of a Non-union.
Description: The existing peer-reviewed literature is inconsistent with respect to the hypothesis that the Oswestry Disability Index (ODI) is affected by a non-union of a lumbar level treated using fusion surgery. The ODI quantifies disability related to low back pain. The ODI is measured on a scale of 0 to 100, with higher scores indicating greater disability. The ODI will be recorded preoperatively and at 12 months following surgery. Each lumbar level will be classified as fused if intervertebral rotation between flexion and extension is < 2 degrees and there is an absence of a discontinuity in bone bridging between vertebrae. The ODI at 12 months, as well as the change in ODI relative to preoperative outcomes will be compared for subjects classified as fused versus not-fused. This test will only be performed for subjects where the stenotic lumbar level was treated using decompression and fusion.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-09

6. Secondary Outcome: Is Leg Pain at 12 Months Following Lumbar Fusion Surgery Dependent on Whether the Treated Level is Fused, With Fusion Defined as Intervertebral Rotation < 2 Degrees and an Absence of Radiographic Signs of a Non-union
Description: The existing peer-reviewed literature is inconsistent with respect to the hypothesis that leg pain assessed using a Numerical Rating Scale (NRS) is affected by a non-union of a lumbar level treated using fusion surgery. Leg pain is measured on a scale of 1 to 10, with higher scores indicating worse leg pain. Leg pain will be recorded preoperatively and at 12 months following surgery. Each lumbar level will be classified as fused if intervertebral rotation between flexion and extension is < 2 degrees and there is an absence of a discontinuity in bone bridging between vertebrae. The leg pain NRS data at 12 months, as well as the change in leg pain relative to preoperative outcomes will be compared for subjects classified as fused versus not-fused. This test will only be performed for subjects where the stenotic lumbar level was treated using decompression and fusion.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Per Protocol: Subject met all inclusion criteria, did not have any exclusion criteria, and had >= 5 deg intervertebrakl rotation at the treatment level at PreOp.
Arm/Group | Per Protocol
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 26/75
Other Adverse Events (participants affected / at risk) | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Per Protocol (N=75)
Recurrent leg pain after decompression surgery (Musculoskeletal and connective tissue disorders) | 1 — Particpant has undergone reoperation to fuse the level where decompression only was the initial surgery chosen in part due to the SPSI metric - investigator assessed this as probably related to use of the SPSI metric
Patient requested two level fusion after 1 level decompression (Musculoskeletal and connective tissue disorders) | 1 — Per the investigators assessment, the adverse event is possibly related to the SPSI metric
Not related to use of SPSI for surgical planning (Musculoskeletal and connective tissue disorders) | 17 — Foot, leg, wrist, infections, and neck/back related issues not related to use of SPSI for surgical planning
Not related to use of SPSI for surgical planning (General disorders) | 7 — Kidney stones, lung embolism, cancer, renal failure

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03754972/Prot_SAP_000.pdf